CLINICAL TRIAL: NCT04193813
Title: Predictors of Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: El-Manial Hospital
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: AF - Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAF
  Interventions: Other: Observational
- Non POAF
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational study

SUMMARY:
There are a wide range of significant epidemiological, clinical, and operative predictors for the development of post-CABG AF including older age, female gender, large LA diameter, higher CHA2DS2-VASc score, valve replacement and postoperative inotropic support. Nevertheless, further large-scale studies are still needed to confirm our findings

DETAILED DESCRIPTION:
We included patients undergoing isolated CABG or CABG with (Aortic and / or Mitral) valve replacement with an age group between 18 and 70 years old.

Patients diagnosed preoperatively with AF or have history of AF, patients with history of existing pre-operative rhythm other than normal sinus rhythm (NSR), patients with impaired systolic function (Ejection fraction (EF) < 30%), patients with end stage renal disease (ESRD) on hemodialysis and patients who refused to participate in the study were excluded from the study.

Sample Size and Sampling: Using PASS program, setting alpha error at 5% and power 80%. Results from previous study Ducceschi et al. (6) showed that left atrial (LA) diameter was an independent factor affecting AF post CABG. Based on this, the needed sample was 123 cases undergoing CABG, including at least 24 patients with dilated LA.

All individuals were monitored for AF during the postoperative ICU stay with continuous ECG (5-leads) monitor, daily 12-lead ECG recording to confirm an episode of AF. AF was considered if P wave was absent before the QRS complex together with irregular ventricular rhythm on the rhythm strips.

Only AF episodes lasting > 5 minutes were counted. In the present study, the following data, as potential predictors of POAF, was collected from every eligible participant; age, sex, smoking and left atrial (LA) diameter based on formal preoperative Trans-thoracic Echocardiography. Serum potassium (K+) level was routinely measured postoperatively on ICU admission and every 2 hours and on demand (if arrhythmia occurs or suspected abnormal potassium level). It was recorded for statistical analysis on admission and every 12 hours and on demand until the patient was discharged.

Serum Magnesium (Mg++) level was measured routinely measured postoperatively on ICU admission and every 24 hours and on demand (if arrhythmia occurs or suspected abnormal magnesium level). It was recorded for statistical study on admission and every 24 hours and on demand until the patient was discharged.

Other parameters such as valve replacement (Aortic and/or Mitral) during the same operative setting, CHA2DS2-VASc score (Congestive heart failure, Hypertension [blood pressure >140/90 mm Hg or treated hypertension on medication], Age ≥75 years, Diabetes mellitus, prior Stroke or transient ischemic attack or thromboembolism, vascular disease, Age 65 to 74 years, Sex category [female sex] ), and post-operative inotropic support usage were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated CABG
* Patients undergoing CABG with (Aortic and / or Mitral) valve replacement
* age group between 18 and 70 years old.

Exclusion Criteria:

* Patients diagnosed preoperatively with AF or have history of AF
* Patients with history of existing pre-operative rhythm other than normal sinus rhythm (NSR)
* Patients with impaired systolic function (Ejection fraction (EF) < 30%)
* Patients with end stage renal disease (ESRD) on hemodialysis
* Patients who refused to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing isolated CABG or CABG with (Aortic and / or Mitral) valve replacement with an age group between 18 and 70 years old.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of POAF | 6 months
  Incidence of POAF 72hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No